CLINICAL TRIAL: NCT05351125
Title: Outcomes Of Interventional Catheterization In Infants Less Than 3 Months With Critical Congenital Heart Disease
Acronym: CHD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: YHAlattar (Other)
Responsible Party: Sponsor-Investigator, YHAlattar, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: catheterization in CHD
Record Dates: First submitted 2022-03-28; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Critical Congenital Heart Disease
MeSH Terms: interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardiac catheterization — catheterization in critical congenital heart disease requiring atrial septostomy or balloon valvuloplastyor PDA stenting

SUMMARY:
Congenital heart disease is the most common birth defect affecting mostly 1 in 100 births(1), critical congenital heart disease is when there is low systemic cardiac output which requires urgent surgery or catheter intervention in the first year of life(2), in low-income countries CCHD is associated with severe high mortality rate due to low health resources, in high-income countries, CCHD is associated with life-long morbidities and a high burden on the health care systems(1-3)

DETAILED DESCRIPTION:
CCHD are classified into three major components:

Left heart obstructions representing 30-40%, complete transposition of the great arteries (mostly 30%), and right heart obstructions (20-30%).

CCHD may present with signs of low cardiac output and hypoperfusion in case of duct dependent systemic circulation or central cyanosis not responding to oxygen in duct dependent pulmonary circulation or two parallel circulations.

Critical congenital heart disease is classified into :

* Congenital heart disease with duct-dependent systemic blood flow (SBF) as:

  1. Critical aortic stenosis
  2. Critical coarctation of the aorta
* Congenital heart disease with duct-dependent pulmonary blood flow (PBF) as:

  1. Critical pulmonary stenosis.
  2. Pulmonary atresia with intact septum.
  3. Severe types of Fallot's tetralogy and pulmonary atresia with VSD.
* Complete transposition of the great arteries (d-TGA) Classified as non-mixture or inadequate shunting at atrial, ventricular, or duct level.

Recent advances in percutaneous neonatal cardiac interventions have improved survival, decreased morbidity, and mortality in newborns with CCHD compared with surgery(4).

Pediatric cardiac catheter interventions have been an established way for the management of CCHD(5).

Balloon atrial septestomy is the standard intervention for patients with D-TGA with ineffective mixing (6), BAS is indicated when there is time lag between diagnosis and arterial switch operation due to transportation and lack of competent surgical team, and it is also indicated in patients with d-TGA with restrictive inter-atrial communication(7).

Ductus arteriosus stenting is used to maintain a reliable source of pulmonary blood flow in patients with duct-dependent cyanotic CHD(5).

The main advantage of ductus arteriosus stenting is the avoidance of surgery and shunt-related side effects , also it promotes significant PA growth compared to a BT shunt alone (8).

Balloon aortic and pulmonary valvuloplasty and balloon coarctation angioplasty are now established procedures for the management of patients with critical pulmonary or aortic stenosis(9).

ELIGIBILITY:
Inclusion Criteria:

* All infants less than 3 months of age with critical congenital heart disease requiring urgent cardiac catheter intervention including

  1. Critical valvular aortic stenosis requiring aortic valvuoplasty.
  2. Pulmonary valvuloplasty for critical valvular pulmonary stenosis.
  3. Pulmonary valvuloplasty in pulmonary atresia with intact IVS after exclusion of RV-dependent coronary circulation.
  4. PDA stenting in duct dependent congenital cyanotic heart disease.
  5. Atrial septostomy to enhance atrial mixing (in transposition of great arteries with restrictive or no inter-atrial communication).
  6. Balloon angioplasty of native coarctation as a palliative measure to stabilize a patient with severely depressed ventricular function.

     Exclusion Criteria:

  <!-- -->

  1. patent ductus arteriosus closure
  2. percutaneous temporary pacemaker implantation for arrhythmia
  3. diagnostic catheterization.
  4. prematurity
  5. low birth weight
  6. bleeding diathesis
  7. sepsis.

Ages: 12 Hours to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants less than 3 months of age with critical congenital heart disease requiring urgent cardiac catheter intervention
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-06-28 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
the effect of cardiac catheter interventions in infants < 3 months with critical congenital heart disease on morbidity and mortality | 6 months post catheterization
  the success rates of urgent cardiac cathetrization
  Type of procedure.
  Procedural outcome:
Delineation of failure of the procedure and its causes | immediate post procedure up to 1montn
  failure of cardiac catheterization with urgent referral to surgery

SECONDARY OUTCOMES:
Complications of trans catheter intervention | 6 month
  Complications
  1. major complications ( Life-threatening complications requiring urgent unplanned surgery or intervention) as cardiac tamponade, cardiac perforation, cardiac valve injury, allergy to anesthesia or drugs, and CPR maneuvers.
  2. (Procedure-related non-life-threatening complications) as: Vascular thrombosis at the site of access, arrhythmia, hypothermia, aggravation of hypoxia, renal insufficiency, and blood loss.
the least and sufficient Procedure time , the radiation time and its side effects | 6 months
  3. Procedure time including (anesthesia time, access time, catheter intervention time, and fluoroscopy time)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakker MK, Bergman JEH, Krikov S, Amar E, Cocchi G, Cragan J, de Walle HEK, Gatt M, Groisman B, Liu S, Nembhard WN, Pierini A, Rissmann A, Chidambarathanu S, Sipek A Jr, Szabova E, Tagliabue G, Tucker D, Mastroiacovo P, Botto LD. Prenatal diagnosis and prevalence of critical congenital heart defects: an international retrospective cohort study. BMJ Open. 2019 Jul 2;9(7):e028139. doi: 10.1136/bmjopen-2018-028139. PMID 31270117
- [Background] Khalil M, Jux C, Rueblinger L, Behrje J, Esmaeili A, Schranz D. Acute therapy of newborns with critical congenital heart disease. Transl Pediatr. 2019 Apr;8(2):114-126. doi: 10.21037/tp.2019.04.06. PMID 31161078
- [Background] Arth AC, Tinker SC, Simeone RM, Ailes EC, Cragan JD, Grosse SD. Inpatient Hospitalization Costs Associated with Birth Defects Among Persons of All Ages - United States, 2013. MMWR Morb Mortal Wkly Rep. 2017 Jan 20;66(2):41-46. doi: 10.15585/mmwr.mm6602a1. PMID 28103210
- [Background] Melekoglu AN, Baspinar O. Transcatheter cardiac interventions in neonates with congenital heart disease: A single centre experience. J Int Med Res. 2019 Feb;47(2):615-625. doi: 10.1177/0300060518806111. Epub 2018 Oct 30. PMID 30373426
- [Background] Alakhfash AA, Jelly A, Almesned A, Alqwaiee A, Almutairi M, Salah S, Hasan M, Almuhaya M, Alnajjar A, Mofeed M, Nasser B. Cardiac Catheterisation Interventions in Neonates and Infants Less Than Three Months. J Saudi Heart Assoc. 2020 May 12;32(2):149-156. doi: 10.37616/2212-5043.1051. eCollection 2020. PMID 33154909
- [Background] Kumar N, Shaikh AS, Kumari V, Patel N. Echocardiography guided bed side balloon atrial septostomy in dextro transposed great arteries (dTGA) with intact ventricular septum (IVS): A resource limited country experience. Pak J Med Sci. 2018 Nov-Dec;34(6):1347-1352. doi: 10.12669/pjms.346.15792. PMID 30559783